CLINICAL TRIAL: NCT03256331
Title: A Phase I, Open-Label, Dose Escalation and Extension Study to Evaluate the Safety, Tolerability and Preliminary Effects of Oral BEL-X-HG in Patients With Advanced Refractory Solid Malignancies
Brief Title: Evaluate the Safety of BEL-X-HG in Advanced Cancer Patients
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: In the light of the on-going COVID-19 pandemic and the resulted difficulty in patient recruitment.
Sponsor: Belx Bio-Pharmaceutical (Taiwan) Corporation (Industry)
Collaborators: A2 Healthcare Taiwan Corporation (Industry)
Responsible Party: Sponsor
Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: BELXHG-SP001
Record Dates: First submitted 2017-08-13; First posted 2017-08-22 (Actual); Last update posted 2020-06-01 (Actual); Status verified 2020-05

CONDITIONS: Advanced Solid Tumors

STUDY DESIGN:
Intervention Model Description: A sequential Dose Escalation Part of four doses following a 3 + 3 design.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- BEL-X-HG (Experimental): 3+3 dose escalation
  Interventions: Drug: BEL-X-HG

INTERVENTIONS:
Drug: BEL-X-HG — This study will be carried out in 2 parts:
  1. A sequential Dose Escalation Part of four doses following a 3 + 3 design where dose escalation will be made based on DLT, for a single cycle (28 days) of BEL-X-HG treatment
  2. A Dose Extension Part of up to 5 cycles (28 days each) at the same dose level (starting dose) of BEL-X-HG treatment
  Escalating dose levels of BEL-X-HG in 5 study cohorts and one modified dose will be as follows:
  * Cohort 1: Dose level 1 - 0.5 g/day (0.25 g, bid)
  * Cohort 2: Dose level 2 - 1.0 g/day (0.5 g, bid)
  * Cohort 3: Dose level 3 - 2.0 g/day (1.0 g, bid)
  * Cohort 4: Dose level 4 - 4.0 g/day (2.0 g, bid) Modified dose level Cohort 5: Dose level 5 - 1.5 g/day (0.75g bid) This re-escalation is allowed only when dose de-escalates from Dose level 3 to Dose level 2, and 1 DLT in 6 evaluable subjects of Dose level 2.

SUMMARY:
This is a Phase I, open-label, uncontrolled, multicenter dose escalation and extension study to determine the maximum tolerated dose (MTD) and dose-limiting toxicity (DLT), to evaluate safety / tolerability and preliminary effects of BEL-X-HG in patients with advanced refractory solid tumors. Dose escalation during the study will be made based on dose-limiting toxicity (DLT).

DETAILED DESCRIPTION:
This study will be carried out in 2 parts:

Part 1: A sequential Dose Escalation Part of four doses following a 3 + 3 design where dose escalation will be made based on dose-limiting toxicity (DLT), for a single cycle (28-days) of BEL-X-HG treatment

Part 2: A Dose Extension Part of up to 5 cycles (28-days each) at the same dose level (starting dose) of BEL-X-HG treatment

Approximately 24-48 eligible subjects with confirmed advanced refractory solid tumors will be enrolled sequentially, in 3 subject cohorts, from the lower to the higher dose cohort into the study. Escalating dose levels of BEL-X-HG in 4 study cohorts and one modified dose will be as follows:

Cohort 1: Dose level 1 - 0.5 g/day (0.25 g, bid)

Cohort 2: Dose level 2 - 1.0 g/day (0.5 g, bid)

Cohort 3: Dose level 3 - 2.0 g/day (1.0 g, bid)

Cohort 4: Dose level 4 - 4.0 g/day (2.0 g, bid)

Modified dose level Cohort 5: Dose level 5 - 1.5 g/day (0.75g bid) This re-escalation is allowed only when dose de-escalates from Dose level 3 to Dose level 2, and 1 DLT in 6 evaluable subjects of Dose level 2.

BEL-X-HG will be administered orally at the assigned dose level for a single cycle consisting of 28 days during the Dose Escalation Part to each subject. Thereafter, if eligible and willing, subjects can continue to Extension Part for 5 more cycles of treatment (each cycle lasting 28 days), at the same assigned dose level of BEL-X-HG treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients of age ≥20 years
2. Pathologically or cytologically confirmed advanced refractory solid tumors for which standard therapy proven to provide clinical benefit does not exist or is no longer effective. It is acceptable for HCC subjects with Child Pugh stage A to confirm diagnosis of the advanced refractory solid tumors by imaging (CT scan).
3. Evaluable disease, at least one measurable target lesion on imaging by RECIST 1.1 (Response Evaluation Criteria in Solid Tumors) criteria.
4. Eastern Cooperative Oncology Group (ECOG) performance score ≤ 2
5. Life expectancy ≥ 3 months
6. Patients able to swallow and retain orally administered medication and does not have any clinically significant gastrointestinal abnormalities that may alter absorption such as malabsorption syndrome or major restriction of the stomach or bowels
7. Laboratory values at screening and baseline (Day 1) of:

   * Absolute neutrophil count (ANC) ≥ 1,500 /mm3
   * Platelets ≥ 75,000 /mm3
   * Hemoglobin (Hb) ≥ 8.5 g/dL
   * Serum creatinine (Cr.) ≤1.5 mg/dL or estimated Glomerular Filtration Rate (eGFR) ≥ 60 mL/min/1.73 m2.

   MDRD Study equation: eGFR = 186 x (SCr)^-1.154 x (age)^0.203 x (0.742 if female) x (1.210 if African American) SCr: serum creatinine in mg/dL; age: in year
8. Patients with primary liver cancer or hepatic metastasis are eligible to enroll, provided that, at screening and baseline (Day 1), the following criteria are met:

   * Total bilirubin (T-Bil) ≤2.0 mg/dL
   * AST and ALT ≤ 5 times the institutional upper limit of normal
   * Child-Pugh Class A; (Score ≤6)
   * Serum albumin ≥2.8 g/dL
9. Patients with a history of esophageal bleeding have varices that have been sclerosed or banded and no bleeding episodes have occurred during the prior 6 months
10. If history of brain metastases treated with radiation therapy, radiation therapy is required to be completed at least 3 months prior to enrolment and metastasis achieve stable disease (SD) since radiation completion
11. Must have recovered from toxicities of previous anti-cancer treatments to NCI-CTCAE version 4.03 grade 1 or lower, except for alopecia
12. Females patient must be either of non-childbearing potential, i.e. surgically sterilized (e.g. tubal ligation, hysterectomy, or ovariectomy) or one year post- menopausal; or, if of childbearing potential, confirmed not pregnant at screening and use of two adequate contraceptive precautions (as per investigator) i.e. condoms plus oral contraceptives or condoms plus endometrial contraceptive devices, during the entire treatment period of this study and for 6 months after exiting from the study
13. Male patients with female partners of childbearing potential must be willing to use a reliable form of contraception (condoms), from screening until 6 months after existing from the study
14. Given signed and dated written informed consent and willing/able to comply with all protocol required visits/procedures

Exclusion Criteria:

1. Primary major surgery < 4 weeks prior to the planned first study treatment day
2. Lactating or pregnant women or plans to be become pregnant
3. Except for alopecia, any drug-related AE from any previous treatments not recovered to NCI-CTCAE version 4.03 grade 1 or lower prior to the planned first study treatment day
4. With active systemic infections, active and clinically significant cardiac diseases, active gastrointestinal diseases, active pulmonary diseases, or medical conditions that may significantly affect adequate absorption of investigational product.
5. Known allergy to BEL-X-HG or its formulation excipients
6. History of autoimmune disease that in the investigator's opinion may be significant to exclude participation in the study
7. Use of any investigational agents or non-registered product within 4 weeks of baseline
8. Known human immunodeficiency virus (HIV) positivity
9. Known hepatitis B virus (HBV) or hepatitis C virus (HCV) carrier who has:

   * serum HBV DNA > 2,000 IU/mL and abnormal ALT (> 5 ULN) (for HBV carrier)
   * abnormal ALT (> 5 ULN) (for HCV carrier)
10. With conditions, judged by the investigator, as unsuitable for the study
11. Mean QTc with Fridericia's correction (QTcF*) greater than 450 ms in screening ECG or history of familial long QT syndrome

    *: Fridericia's formula:
12. Any cancer-directed therapy (chemotherapy, radiotherapy, biological or immunotherapy, etc.) within 4 weeks or 5 half-lives, (whichever is shorter) of baseline

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2017-06-21 (Actual); Primary Completion 2020-03-30 (Actual); Study Completion 2020-03-30 (Actual)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (MTD) | 28 days (first treatment cycle of every subjects)
  The prior dose level below the dose level at which ≥2/3 or ≥2/6 subjects suffer dose-limiting toxicity (DLT).

SECONDARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events | up to 168 days (up to 6 cycles of each enrolled subjects)
  Incidence of Adverse Events (AEs) and Serious Adverse Events (SAEs)
Tumor response per Response Evaluation Criteria in Solid Tumors (RECIST) | up to 168 days (up to 6 cycles of each enrolled subjects)
  Tumor response per Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1
Oxidative stress | up to 168 days (up to 6 cycles of each enrolled subjects)
  Oxidative stress
nutritional status | up to 168 days (up to 6 cycles of each enrolled subjects)
  serum prealbumin, triglyceride, and total cholesterol
immunological status | up to 168 days (up to 6 cycles of each enrolled subjects)
  TNF-alpha, IL-1, IL-2, IL-4, and IL-6
cachexia status | up to 168 days (up to 6 cycles of each enrolled subjects)
  fast blood glucose, C-reactive protein, and testosteron
Quality of life (QoL) of patients with advanced refractory solid tumors | up to 168 days (up to 6 cycles of each enrolled subjects)
  SF-36 Quality of Life (QoL) Questionnaire
liver function | up to 168 days (up to 6 cycles of each enrolled subjects)
  serum AST, ALT, AKP, albumin, gamma-GT, ferritin, PT/INR and APRI

CONTACTS AND LOCATIONS:
Overall Officials: Chia-Chi Lin, MD, PhD, Principal Investigator — National Taiwan University Hospital
Locations (2):
- Taiwan (2):
  - National Cheng Kung University Hospital, Tainan
  - National Taiwan University Hospital, Taipei

IPD SHARING:
Plan to Share IPD: No